CLINICAL TRIAL: NCT05316220
Title: A Randomized, Double-blind Study to Assess the Safety and Efficacy of Mesalamine Delayed-release Capsules in Children Aged 5 to 17 Years for the Maintenance of Remission of Ulcerative Colitis
Brief Title: A Study to Assess Adverse Events and Change in Disease Condition of Mesalamine Capsules in Children Aged 5 to 17 Years With Ulcerative Colitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-517
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis (UC); Mesalamine; Delzicol; AGN-226474
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesalamine Dose A (Experimental): Participants will receive mesalamine Dose A twice daily for 26 weeks.
  Interventions: Drug: Mesalamine
- Mesalamine Dose B (Experimental): Participants will receive mesalamine Dose B twice daily for 26 weeks.
  Interventions: Drug: Mesalamine; Drug: Placebo

INTERVENTIONS:
Drug: Mesalamine — Oral Capsules
  Other Names: Delzicol
Drug: Placebo — Oral Capsule
  Arms: Mesalamine Dose B

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease (IBD) characterized by diffuse, continuous inflammation of the colon. This study will assess how safe and effective mesalamine delayed-release capsules are in treating pediatric participants with UC. Adverse events and change in disease activity will be assessed.

Delzicol (Mesalamine) is an approved drug being developed for the treatment of Ulcerative Colitis (UC). Study doctors put the participants in 1 of 2 groups, called treatment arms. Each group receives a different treatment. Around 80 Pediatric participants aged 5 to 17 years with a diagnosis of UC will be enrolled in approximately 45 sites in the United States.

Participants will receive oral mesalamine capsules twice daily for 26 weeks and followed for 30 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

- Documented history of Ulcerative Colitis (UC) who have been successfully maintained in remission for at least 30 days prior to the screening visit and are on a stable dose of mesalamine or 5-aminosalicylic acid equivalent.

Exclusion Criteria:

- Abnormal and clinically significant results according to the investigator or designee, on physical examination, medical history, electrocardiogram (ECG), hematology, clinical chemistry, or urinalysis.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-19 (Estimated); Study Completion 2026-07-19 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Maintaining Clinical Remission Responder Status Based on the modified Mayo Score (mMS) | Week 26
  Clinical remission responder based on the mMS is defined as Endoscopy subscore = 0 or 1, AND Rectal bleeding subscore = 0, AND Stool frequency subscore <= 1.

SECONDARY OUTCOMES:
Percentage of Participants Maintaining Endoscopic Remission Responder Status Based on the mMS | Week 26
  Endoscopic remission responder based on the mMS is defined as Endoscopy subscore = 0 or 1.
Percentage of Participants Maintaining Symptomatic Remission Responder Status Based on the mMS | Week 26
  Symptomatic remission responder based on the mMS s defined as Rectal bleeding subscore = 0 AND Stool frequency subscore <= 1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (8):
  - Childrens National /ID# 243379, Washington D.C., District of Columbia
  - Angel Kids Pediatrics /ID# 244874, Jacksonville, Florida
  - Treken Primary Care /ID# 241302, Atlanta, Georgia
  - Eagle Clinical Research /ID# 242045, Chicago, Illinois
  - Virgo Carter Pediatrics /ID# 241556, Silver Spring, Maryland
  - UH Cleveland Medical Center /ID# 243375, Cleveland, Ohio
  - Children's Hospital Oklahoma /ID# 242614, Oklahoma City, Oklahoma
  - Carilion Medical Center /ID# 244398, Roanoke, Virginia
- Puerto Rico (2):
  - San Juan Bautista School of Medicine /ID# 243377, Caguas
  - Centro de Investigaciones Clinicas San Jorge Children's and Women's Hospital /ID# 244595, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com